CLINICAL TRIAL: NCT04226911
Title: Sweeteners and Sweetness Enhancers: Prolonged Effects on Health, Obesity and Safety
Acronym: SWEET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Birgitte Raben (Other)
Collaborators: Harokopio University (Other); University of Navarra (Other); University of Liverpool (Other); Maastricht University (Other); University of Leeds (Other); Wageningen University (Other); European Clinical Research Infrastructure Network (Other); University of Surrey (Other); Bioiatriki Idiotiko Polyiatreio Iatpikh Anonymos Etairia (Unknown); NetUnion SARL (Unknown); Pectolite GMBH (Unknown)
Responsible Party: Sponsor-Investigator, Anne Birgitte Raben, Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SWEET WP3
Record Dates: First submitted 2019-12-18; First posted 2020-01-13 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Sugars

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sweeteners and sweetness enhancers (S&SEs) (Experimental): Healthy diet < 10 energy % (E%) sugar, foods and drinks with S&SEs allowed.
  Interventions: Behavioral: S&SEs
- Sugar group (Active Comparator): Healthy diet, < 10 E% sugar, foods and drinks with S&SEs not allowed.
  Interventions: Behavioral: Sugar

INTERVENTIONS:
Behavioral: S&SEs — S&SEs:
  As many sugar-containing products in the diet as possible should be replaced with S&SE-containing products.
  To ensure that a certain amount of S&SE products is consumed every day, a fixed minimum amount of units for each individual is planned.
  Arms: Sweeteners and sweetness enhancers (S&SEs)
Behavioral: Sugar — Sugar group:
  In the sugar group it is allowed to consume up to a certain number of units of sugar-containing products each day, corresponding to < 10 E% added sugar.
  The sugar group is not allowed to consume any S&SE products.
  Arms: Sugar group

SUMMARY:
The aim of this randomised controlled trial (RCT) is to investigate if prolonged consumption of sweetener and sweetness enhancers (S&SEs) within a healthy diet approach will improve weight loss maintenance and obesity related risk factors, and affect safety markers, compared to sugar.

We hypothesize, that:

* Prolonged use of S&SEs in beverages and food matrices will result in improved body weight control because S&SEs will increase palatability of the diet and thereby increase compliance to the recommendations for a healthy diet.
* There will be no safety concerns using S&SEs in the long term.

Overweight/obese adults and families where at least one adult (both gender) and one child (both gender) are overweight/obese will be recruited. The majority of measurements will only be conducted in the adult population and some measurement will only be done in sub-groups. The intervention will be performed in four countries: Denmark, Greece, Spain and the Netherlands.

The goal is approximately 370 participants - 330 adults (18-65 years of age) and 40 children (6-12 years of age) - will be recruited for the study. All adult participants are first treated by a low energy diet (LED) for 2 months with the aim to reduce body weight (minimum 5% weight loss (WL)), whereas children are treated separately with a conventional weight maintenance (WM) diet, without a specific aim for absolute WL.

The participants - both adults and families - are randomized into two different diet interventions for 10 months with or without inclusion of S&SEs products (foods and drinks). For adults, this period aims at preventing weight re-gain and for children maintaining body mass index (BMI)-for-age. The participants will receive food exchange lists and will be guided by dieticians. The randomization will be stratified by age, sex and BMI. Adults (not participating with children) belonging to the same household and all members of a family will be assigned the same intervention - the randomization will here solely be based on the oldest adult in the family/household.

The adult participants are weighed at months 0, 0.5 and 1, and if needed at month 1.5. They are supervised during the WL period at months 0 and 1, and if needed at months 0.5 and 1.5, and throughout the WM period at months 2, 4, 6, 9 and 12. Children will follow a similar, but less strict time schedule (their participation is preferred but not required for all dietician meetings).

The main assessment points are the clinical investigation days (CIDs) at month 0 (baseline, start of the WL period), 2 (end of the WL period/start of randomized intervention), 6 (6 months from baseline) and 12 (1 year from baseline).

ELIGIBILITY:
Inclusion criteria for adults:

* Age: 18-65 years.
* BMI: ≥25.0 kg/m2 (no upper limit). For women: Use of contraceptive methods and not wishing/planning to become pregnant in the 1 year of the intervention study.
* Regular consumption of sugar-containing/sugar-sweetened products.
* Able to participate in CIDs and dietician meetings during normal working hours.
* Motivation and willingness to be randomized to any of the two groups and to do the best to follow the given protocol.

Inclusion criteria for children:

* Age: 6-12 years.
* BMI-for-age: >85th percentile (no upper limit).
* Able to participate in CIDs during normal working hours.
* Motivation and willingness to be randomized to any of the two groups and to do the best to follow the given protocol.

Exclusion criteria for adults:

* Weight change (increase or decrease) >5% during the past 2 months prior to the study.
* Surgical treatment of obesity.
* Blood donation < 3 month prior to study.
* Change in smoking habits during the last month. Smoking is allowed provided subjects have not recently changed habits. However, smoking status is monitored throughout the study and used as a confounding variable.
* Regularly drinking >21 alcoholic units per week (men), or >14 alcoholic units/week (women).
* Intensive physical training (>10 hours of per week).
* Self-reported eating disorders.
* Intolerance and allergies expected to interfere with the study.
* Self-reported drug abuse within the previous 12 months.
* Night- or shift work that ends later than 11 PM.
* For women: Pregnancy, lactation.
* Persons who do not have access to either (mobile) phone or internet (this is necessary when being contacted by the study personnel during the study).
* Insufficient communication with national language.
* Inability, physically or mentally, to comply with the procedures required by the study protocol as evaluated by the daily study manager, site-PI, PI or clinical responsible
* Participant's general condition contraindicates continuing the study as evaluated by the daily study manager, site-PI, PI or clinical responsible.
* Simultaneous participation in other clinical intervention studies.

Medical conditions as known by the persons:

* Diagnosed diabetes mellitus.
* Medical history of CVD (e.g. current angina; myocardial infarction or stroke within the past 6 months; heart failure; symptomatic peripheral vascular disease).
* Systolic blood pressure above 160 mmHg and/or diastolic blood pressure above 100 mmHg (measured at screening) whether on or off treatment for hypertension.
* Significant liver disease, e.g. cirrhosis (fatty liver disease allowed).
* Malignancy which is currently active or in remission for less than five years after last treatment (local basal and squamous cell skin cancer allowed).
* Active inflammatory bowel disease, celiac disease, chronic pancreatitis or other disorder potentially causing malabsorption.
* Thyroid diseases, except those on Levothyroxine treatment of hypothyroidism if the person has been on a stable dose for at least 3 months.
* Psychiatric illness (e.g. major depression, bipolar disorders).

Medication:

* Use currently or within the previous 3 months of prescription or over the counter medication that has the potential of affecting body weight incl. food supplements. Except: low dose antidepressants if they, in the judgement of the daily study manager, site-PI, PI or clinical responsible, do not affect weight or participation to the study protocol. Levothyroxine for treatment of hypothyroidism is allowed if the person has been on a stable dose for at least 3 months.
* Cholesterol or blood pressure lowering medication, if the dose has changed during the last 3 months (i.e. the medication is allowed if the participant has been on a stable dose for at least 3 months).

Laboratory screening:

If all of the above criteria are satisfied, the adult participant is eligible for a laboratory screening. A blood sample is collected and immediately analysed for glucose and haemoglobin concentrations (Haemocue).

* Glucose ≥ 7.0 mmol/L.
* Haemoglobin concentration below local laboratory reference values (i.e. anaemia).
* Or any other significant abnormality on these tests which in the investigators opinion may be clinically significant and require further assessment.

After WL period (CID2, Month 2):

Failure to reach at least 5% weight reduction during the WL period (Months 0-2). This leads to exclusion from the WM intervention

Exclusion criteria for children:

* Intensive physical training (>10 hours of per week).
* Self-reported eating disorders.
* Intolerance and allergies expected to interfere with the study.
* Insufficient communication with national language.
* Inability, physically or mentally, to comply with the procedures required by the study protocol as evaluated by the daily study manager, site-PI, PI or clinical responsible.
* Subject's general condition contraindicates continuing the study as evaluated by the daily study manager, principal investigator or clinical responsible.
* Simultaneous participation in other clinical intervention studies.

Medical conditions as known by the child and the representative adult:

* Diagnosed diabetes mellitus.
* Other diseases that may influence the study outcomes as evaluated by the daily study manager, site-PI, PI or clinical responsible.

Medication:

* Use currently or within the previous 3 months of prescription or over the counter medication that has the potential of affecting body weight.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Change in body weight (adults) | Up to 1 year.
  Efficacy: Change in body weight will be measured by a calibrated digital scale.
Changes in gut microbiota composition (adults) | Up to 1 year.
  Safety: Change in gut microbiota associated with impaired health (e.g. change in microbial beta-diversity and composition) will be measured by fecal samples.

SECONDARY OUTCOMES:
Change in BMI-for-age z-score (children) | Up to 1 year.
  Efficacy: Efficacy: BMI-for-age z-score will be calculated based on the childrens weight and height using WHO AnthroPlus.
Changes in waist and hip circumferences (adults and children) | Up to 1 year.
  Efficacy: Changes in waist and hip circumferences will be measured with a non-elastic tape.
Change in body composition (adults and children) | Up to 1 year.
  Efficacy: Body composition will be measured using Dual X-rays. Children are not DXA scanned at UM.
Change in blood pressure and heart rate (adults and children) | Up to 1 year.
  Efficacy: Change in blood pressure will be measured by an automatic device on the right arm.
Change in glucose (adults and children) | Up to 1 year.
  Efficacy: Change in glucose will be measured by fasting blood samples.
Change in hemoglobin A1c (adults and children) | Up to 1 year.
  Efficacy: Change in hemoglobin A1c will be measured by fasting blood samples.
Change in alanine aminotransferase (ALT) (adults and children) | Up to 1 year.
  Efficacy: Change in ALT will be measured by fasting blood samples.
Change in aspartate aminotransferase (AST) (adults and children) | Up to 1 year.
  Efficacy: Change in AST will be measured by fasting blood samples.
Change in insulinemia (adults and children) | Up to 1 year.
  Efficacy: Change in insulinemia (insulin) will be measured by fasting blood samples.
Change in lipidemia (adults and children) | Up to 1 year.
  Efficacy: Change in lipidemia (total cholesterol, high-density cholesterol, low-density cholesterol, triglycerides) will be measured by fasting blood samples.
Change C-reactive protein (CPR) (adults and children) | Up to 1 year.
  Efficacy: Change in CPR will be measured by fasting blood samples.
Allergenicity by serum immunoglobulin level (adults and children) | Up to 1 year.
  Safety: To assess allergenicity serum immunoglobulin levels will be measured by fasting blood samples.
Allergenicity by a skin prick test (adults) | Up to 1 year.
  Safety: To assess allergenicity a skin prick test will be performed.
Allergenicity by a questionnaire (adults and children) | Up to 1 year.
  Safety: To assess allergenicity a questionnaire will be completed.
Concomitant medication (adults and children) | Up to 1 year.
  Safety: Concomitant medication will be reported in a case report from designed for the purpose.
Adverse events (adults and children) | Up to 1 year.
  Safety: Adverse events will be reported in a case report form designed for the purpose e.g. headache, constipation ect.
Change in liver fat and lipid composition (adults) | Up to 1 year.
  Safety: Change in liver fat and lipid composition will be measured by magnet resonans (MR) scans in a sub-group (UM).
Change in ghrelin (adults) | Up to 1 year.
  Efficacy: Change in ghrelin will be measured in a sub-group by fasting blood samples (UCPH, UM).
Change in cholecystokinin (adults) | Up to 1 year.
  Efficacy: Change in cholecystokinin will be measured in a sub-group by fasting blood samples (UCPH, UM).
Change in glucagon-like peptide-1 (GLP-1) (adults) | Up to 1 year.
  Efficacy: Change in GLP-1 will be measured in a sub-group by fasting blood samples (UCPH, UM).
Change in FGF21 (adults) | Up to 1 year.
  Efficacy: Change in FGF21 will be measured in a sub-group by fasting blood samples (UCPH).
Changes in gut microbiota composition (children) | Up to 1 year.
  Safety: Change in gut microbiota associated with impaired health (e.g. change in microbial beta-diversity and composition) will be measured by fecal samples in a sub-group (UM)
Markers of adipogenesis (adults) | Up to 1 year.
  Safety: Markers of adipogenesis will be measured by a adipose tissue biopsy (needle biopsy) in a sub-group (UM).
Lipolysis (adults) | Up to 1 year.
  Safety: Markers of lipolysis will be measured by a adipose tissue biopsy (needle biopsy) in a sub-group (UM).
Fat cell size (adults) | Up to 1 year.
  Safety: Change in fat cell size will be measured by a adipose tissue biopsy (needle biopsy) in a sub-group (UM).
Inflammation markers (adults) | Up to 1 year.
  Safety: Change in inflammation markers will be measured by a adipose tissue biopsy (needle biopsy) in a sub-group (UM).
Insulin sensitivity (adults) | Up to 1 year.
  Efficacy: Insulin sensitivity will be measured by a 7-point oral glucose tolerance test (OGTT) in a sub-study (UM).
Glucose tolerance (adults) | Up to 1 year.
  Efficacy: Glucose tolerance will be measured by a 7-step oral glucose tolerance test (OGTT) in a sub-study (UM).
Changes in gut-microbial composition in response to specific S&SEs in vitro (adults) | Only baseline feces samples will be used
  Safety: Changes in gut-microbial composition will be measured in the TIM-2 model of the human colon in response to specific S&SEs in a sub-group (UM).
Changes in gut-microbial functionality in response to S&SEs in vitro (adults) | Up to 1 year.
  Safety: Changes in gut-microbial functionality (metabolite production) will be assessed in the TIM-2 model of the human colon in response to specific S&SEs in a sub-group (UM).
Baseline and postprandial energy expenditure (adults) | Up to 6 months.
  Efficacy: Energy expenditure will be measured in a sub-group by the ventilated hood system - a sub-study at UCPH.
Baseline and postprandial substrate oxidation (adults) | Up to 6 months.
  Efficacy: The substrate oxidation will be measured only in a sub-group of adults by the ventilated hood system - a sub-study at UCPH.
Baseline and postprandial appetite (adults) | Up to 6 months.
  Efficacy: Appetite will be measured only in a sub-group by visual analog scales and acute energy intake - a sub-study at UCPH.
Baseline and postprandial blood samples (adults) | Up to 6 months.
  Efficacy: Blood samples will be taken in a small group of the participants in the sub-study at UCPH.

OTHER OUTCOMES:
Food preferences (adults and children) | Up to 1 year.
  Neuro-behavioral: Food preferences will be measured by questionnaires.
Perception of S&SEs (adults) | Up to 1 year.
  Neuro-behavioral: Perception of S&SEs will be measured by a questionnaire.
Cravings (adults) | Up to 1 year.
  Neuro-behavioral: Cravings will be measured by questionnaires.
Subjective appetite sensation (adults) | Up to 1 year.
  Neuro-behavioral: Subjective appetite sensation will be measured by visual analogue scales (VAS).
Perception and evaluation of the weight maintenance intervention (adults) | Up to 1 year.
  Neuro-behavioral: Perception and evaluation of the weight maintenance intervention will be measured by questionnaires.
Dietary restraint and disinhibition (adults and children) | Up to 1 year.
  Neuro-behavioral: Dietary restraint and disinhibition will be measured by a questionnaire.
Dietary intake (adults and children) | Up to 1 year.
  Dietary intake is measured by dietary records.
Biomarkers (adults) | Up to 1 year.
  Biomarkers is measured by urine samples.
Physical activity (adults and children) | Up to 1 year.
  Physical activity will be monitored in detail by accelerometers in a sub-group of the adults and by a questionnare for all participants.
Brain reward activity (adults) | Up to 1 year.
  Assessment of brain reward activity is measured by functional Magnetic Resonance Imaging (fMRI) in a sub-group - a sub-study at UM.
Puberty (children) | Up to 1 year.
  Pubertal maturation will be assessed by a self-assessment questionnare.

CONTACTS AND LOCATIONS:
Locations (4):
- Department of Nutrition, Exercise and Sports, Frederiksberg, Denmark
- Harokopio University, Kallithea-Athens, Greece
- University of Maastricht, Maastricht, Netherlands
- University of Navarra, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All data will be collected in a central DataHub at University of Copenhagen. First, the pseudo-anonymised individual participant data (IPD) are to be shared between (WP3-) relevant SWEET partners within the SWEET consortium via a data processor agreement (DPA). Second, the pseudo-anonymised IPD will be made available upon request before 2032 via a data sharing contract. Third, from 2032 (10 years after LPLV) fully anonymised data can be transferred."
Supporting Information: Study Protocol
Time Frame: See above in the plan description.
Access Criteria: See above in the plan description.

REFERENCES:
- [Derived] Pang MD, Kjolbaek L, Bastings JJAJ, Andersen SSH, Umanets A, Sost MM, Navas-Carretero S, Reppas K, Finlayson G, Hodgkins CE, Del Alamo M, Lam T, Moshoyiannis H, Feskens EJM, Adam TCM, Goossens GH, Halford JCG, Harrold JA, Manios Y, Martinez JA, Blaak EE, Raben A. Effect of sweeteners and sweetness enhancers on weight management and gut microbiota composition in individuals with overweight or obesity: the SWEET study. Nat Metab. 2025 Oct;7(10):2083-2098. doi: 10.1038/s42255-025-01381-z. Epub 2025 Oct 7. PMID 41057614
- [Derived] Pang MD, Bastings JJAJ, Op den Kamp-Bruls YMH, Harrold JA, Kjolbaek L, Halford JCG, Adam TCM, Raben A, Schrauwen-Hinderling VB, Goossens GH, Blaak EE. The effect of weight loss on whole-body and tissue-specific insulin sensitivity and hepatic lipid content and composition: SWEET substudy. Obesity (Silver Spring). 2023 Jul;31(7):1745-1754. doi: 10.1002/oby.23773. PMID 37368517
- [Derived] Kjolbaek L, Manios Y, Blaak EE, Martinez JA, Feskens EJM, Finlayson G, Andersen SSH, Reppas K, Navas-Carretero S, Adam TC, Hodgkins CE, Del Alamo M, Lam T, Moshoyiannis H, Halford JCG, Harrold JA, Raben A. Protocol for a multicentre, parallel, randomised, controlled trial on the effect of sweeteners and sweetness enhancers on health, obesity and safety in overweight adults and children: the SWEET project. BMJ Open. 2022 Oct 12;12(10):e061075. doi: 10.1136/bmjopen-2022-061075. PMID 36223962